CLINICAL TRIAL: NCT01844882
Title: The Effects of Dietary Fiber on Uremic Retention Solutes in CKD: A Systematic Review and Meta-analysis
Brief Title: The Effects of Dietary Fiber in CKD: A Systematic Review and Meta-analysis
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: SMH-CKD-2013
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Kidney Disease
Keywords: The effects; dietary; fiber; kidney function; CKD patients
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease

SUMMARY:
Chronic kidney disease (CKD) is a debilitating condition in which there is a gradual decline of renal function associated with increased overall mortality. Most dietary guidelines for CKD focus on limiting protein intake (nitrogen) and high phosphorus-containing foods. However, increasing dietary fiber has been proposed to increase fecal nitrogen excretion which may ameliorate the progress of CKD. We therefore plan to conduct a systematic review and meta-analysis on clinical trials to assess the effect of fiber on urea and creatinine as classical markers of a state of uremia in individuals with CKD. We hypothesize that increasing fiber intakes will improve urea and creatinine levels in individuals with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Dietary trials in humans
* Randomized treatment allocation
* Suitable control (low fiber)
* viable endpoint data

Exclusion Criteria:

* Non-human studies
* Nonrandomized treatment allocation
* Lack of a suitable control (high protein)
* no viable endpoint data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Chronic Kidney Disease (CKD)
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Creatinine | 1.5 years
urea | 1.5 years

SECONDARY OUTCOMES:
Phosphorus | 1.5 years

REFERENCES:
- [Derived] Chiavaroli L, Mirrahimi A, Sievenpiper JL, Jenkins DJ, Darling PB. Dietary fiber effects in chronic kidney disease: a systematic review and meta-analysis of controlled feeding trials. Eur J Clin Nutr. 2015 Jul;69(7):761-8. doi: 10.1038/ejcn.2014.237. Epub 2014 Nov 12. PMID 25387901